CLINICAL TRIAL: NCT05466929
Title: Supporting Mental Health in Underserved Youth: Engagement With Digital Mental Health Technologies in Pediatric Primary Care
Brief Title: Engagement With Digital Mental Health (DMH) Technologies in Pediatric Primary Care
Acronym: TeACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K08MH125069 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-20 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Mental Health
Keywords: Digital Mental Health Technology; Digital Mental Health; Mental Health Disorders; Mental Health Wellness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Intervention group (TeACH System psychoeducation and recommendations) and control group (evidence-based online educational materials)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TeACH System Resources (Experimental): Patients who screen positive for anxiety will receive stakeholder-informed feedback and resources (i.e., psychoeducation and mental health recommendations).
  Interventions: Behavioral: TeACH System Resources
- Evidence-based Resources (No Intervention): Patients who screen positive for anxiety will receive a link to a webpage providing psychoeducation about anxiety and possible treatment options.

INTERVENTIONS:
Behavioral: TeACH System Resources — Patients who screen positive for anxiety will receive psychoeducation and mental health recommendations (e.g., evidence-based apps) selected for use with the TeACH System through a collaborative, stakeholder-engaged approach completed in phases 1 and 2 of this project.
  Arms: TeACH System Resources

SUMMARY:
The goal of this study is to use and adapt existing digital mental health technologies to advance the engagement, assessment, detection, treatment, and delivery of services for pediatric mental health in families from underserved communities.

DETAILED DESCRIPTION:
The goal of this study is to use and adapt existing digital mental health technologies to advance the engagement, assessment, detection, treatment, and delivery of services for pediatric mental health. Specifically, user-centered design methodologies and an implementation science framework will be used to guide the development and implementation of the Teen Assess, Check, and Heal (TeACH) System into a pediatric primary care clinic serving teens and families from underserved communities.

Study objectives include:

1. Collaborating with underserved teens and their parents to identify strategies to target top barriers to engagement as well as top ethical concerns and requirements for cultural relevance, usability, and usefulness of the TeACH System (Phase 1)
2. Refining the plan for implementing the TeACH System through observations, interviews, and co-design workshops with pediatric primary care pediatricians and staff (Phase 2), and
3. Implementing the TeACH System into a primary care clinics and evaluating it in a randomized trial. (Phase 3)

The team will measure engagement outcomes and satisfaction with the TeACH System

ELIGIBILITY:
Inclusion Criteria:

* Are receiving care at specified Rush University Health System and University of Illinois at Chicago Pediatric Primary Care locations
* Are between 13-17 years of age
* Are able to speak and read in English
* Symptoms of anxiety disorder

Exclusion Criteria:

* Absence of the above inclusion criteria.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 365 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-11-06 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Anxiety Understanding: Baseline | Administered following assent (in case of participant attrition through the interaction)
  1 item (Likert Scale); We will ask participants to rate their understanding of anxiety on a Likert scale (1-5; 1 being "Not at All" and 5 being "Completely"). Specifically: "I understand what anxiety is."
Anxiety Understanding: Post Interaction | Administered immediately after receiving randomized feedback/resources
  1 item (Likert Scale); We will ask participants to rate their understanding of anxiety on a Likert scale (1-5; 1 being "Not at All" and 5 being "Completely"). Specifically: "I understand what anxiety is."
Anxiety Understanding: Maintenance | Administered one week after interaction with TeACH System
  1 item (Likert Scale); We will ask participants to rate their understanding of anxiety on a Likert scale (1-5; 1 being "Not at All" and 5 being "Completely"). Specifically: "I understand what anxiety is."
Confidence to Act: Baseline | Administered following assent (in case of participant attrition through the interaction)
  1 item (Likert Scale); We will ask participants to rate how confident they feel to take action to help their anxiety symptoms on a Likert scale (1-5; 1 being "Not at All" to 5 being "Completely"). Specifically: "I feel confident I can do something if I feel anxiety."
Confidence to Act: Post Interaction | Administered immediately after receiving randomized feedback/resources
  1 item (Likert Scale); We will ask participants to rate how confident they feel to take action to help their anxiety symptoms on a Likert scale (1-5; 1 being "Not at All" to 5 being "Completely"). Specifically: "I feel confident I can do something if I feel anxiety."
Confidence to Act: Maintenance | Administered one week after interaction with TeACH System
  1 item (Likert Scale); We will ask participants to rate how confident they feel to take action to help their anxiety symptoms on a Likert scale (1-5; 1 being "Not at All" to 5 being "Completely"). Specifically: "I feel confident I can do something if I feel anxiety."
Likelihood of using DMH for Anxiety: Baseline | Administered following assent (in case of participant attrition through the interaction)
  1 item (Likert Scale); We will ask participants to rate how likely they are to use digital mental health tools for their anxiety on a Likert scale (1-5; 1 being "Never" to 5 being "Absolutely"). Specifically: "If I feel anxiety, I would use a digital tool to help (app, website, reel/video)."
Likelihood of using DMH for Anxiety: Post Interaction | Administered immediately after receiving randomized feedback/resources
  1 item (Likert Scale); We will ask participants to rate how likely they are to use digital mental health tools for their anxiety on a Likert scale (1-5; 1 being "Never" to 5 being "Absolutely"). Specifically: "If I feel anxiety, I would use a digital tool to help (app, website, reel/video)."
Likelihood of using DMH for Anxiety: Maintenance | Administered one week after interaction with TeACH System
  1 item (Likert Scale); We will ask participants to rate how likely they are to use digital mental health tools for their anxiety on a Likert scale (1-5; 1 being "Never" to 5 being "Absolutely"). Specifically: "If I feel anxiety, I would use a digital tool to help (app, website, reel/video)."
DMH use for Anxiety: Baseline | Administered following assent (in case of participant attrition through the interaction)
  1 item (Yes/No/Unsure); We will ask participants to report if they have used digital mental health tools for their anxiety symptoms. Specifically: "I have used a digital tool to help with anxiety (app, website, reel/video)."
DMH use for Anxiety: Post Interaction | Administered immediately after receiving randomized feedback/resources
  1 item (Yes/No/Unsure); We will ask participants to report if they have used digital mental health tools for their anxiety symptoms. Specifically: "I have used a digital tool to help with anxiety (app, website, reel/video)."
DMH use for Anxiety: Maintenance, Change in DMH Use Following TeACH System Interaction | Administered one week after interaction with TeACH System
  1 item (Yes/No/Unsure); We will ask participants to report if they have used digital mental health tools for their anxiety symptoms. Specifically: "I have used a digital tool to help with anxiety (app, website, reel/video)."
Enrollment | Through study completion, an average of once per year.
  We will track the number of teens who use the TeACH System during implementation phases and will compare this to the number of teens who were eligible but did not use the system.

SECONDARY OUTCOMES:
Kiddie-Computerized Adaptive Tests (K-CAT) Anxiety Module | Administered immediately after initiating use of the TeACH System; teen participants complete only once.
  <1 minute to complete; Uses item response theory to pull from a large question item bank to accurately diagnose anxiety symptom severity.
After-Scenario Questionnaire (ASQ): Post Interaction | Administered immediately after receiving randomized feedback/resources from TeACH System
  3-item tool with seven response options (1-Strongly Disagree to 7-Strongly Agree) to assess satisfaction
After-Scenario Questionnaire (ASQ): Maintenance | Administered one week after interaction with TeACH System
  3-item tool with seven response options (1-Strongly Disagree to 7-Strongly Agree) to assess satisfaction

OTHER OUTCOMES:
Demographics | Administered immediately after initiating use of the TeACH System; teen participants complete only once.
  Name, date of birth, ethnicity, race, pronouns, gender, preferred language, reason for visiting primary care today, preferred channel of contact (i.e., text or email for follow-up)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois

REFERENCES:
- [Derived] Stiles-Shields C, Bobadilla G, Reyes K, Gustafson EL, Lowther M, Smith DL, Frisbie C, Antognini C, Dyer G, MacCarthy R, Martinengo N, Morris G, Touranachun A, Wilkens KM, Julion WA, Karnik NS. Digital Mental Health Screening, Feedback, and Referral System for Teens With Socially Complex Needs: Protocol for a Randomized Controlled Trial Integrating the Teen Assess, Check, and Heal System into Pediatric Primary Care. JMIR Res Protoc. 2025 Feb 18;14:e65245. doi: 10.2196/65245. PMID 39965196